CLINICAL TRIAL: NCT04580615
Title: Anonymized Data Collection From the CardiacSense1 and Other Modalities for the Purpose of Developing a System for Monitoring of Respiratory Rate
Brief Title: Data Collection From the CardiacSense1 and Other Modalities for Developing a System for Monitoring of Respiratory Rate
Acronym: RRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CL00450
Record Dates: First submitted 2020-04-16; First posted 2020-10-08 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Disease
Keywords: Respiratory rate
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inpatients subjects (Experimental): Inpatients subjects diagnosed with a Respiratory disease/impairment or subjects with no known Respiratory disease/impairment
  Interventions: Device: CardiacSense1 and capnograph Respiratory rate measurement

INTERVENTIONS:
Device: CardiacSense1 and capnograph Respiratory rate measurement — Inpatients Subjects with respiratory disease/impairment and Inpatients Subjects with no known respiratory disease/impairment will be measured simultaneously with both CardiacSense1 and capnograph for at least 30 minutes up to 24 hours. During this time capnograph data will be recorded in parallel to CardiacSense1.

SUMMARY:
Collect data from the CardiacSense1's sensors and Capnograph, for the purpose of developing a wearable system for monitoring of Respiratory Rate (RR) in patients while at hospital

DETAILED DESCRIPTION:
Hospitalized subjects, diagnosed with a Respiratory disease or subjects with no known Respiratory disease will be will be connected simultaneously to CardiacSense watch and Capnograph for a duration of at least 30 minutes and up to 24 hours in order to collect data for the purpose of developing a wearable system for monitoring of Respiratory Rate (RR) by the CardiacSense watch.

The CardiacSense1 is a wrist worn device designed to detect atrial fibrillation. CardiacSense1 senses the radial artery inflation and deflation and together with a PPG sensors give an ultimate performance that is superior to PPG only.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen (18) year and above
* Diagnosed with Respiratory disease/impairment or without any known Respiratory disease/impairment
* Ability and willingness to sign an informed consent form

Exclusion Criteria:

* Subjects who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the subject's participation in this study
* Patients with significant co morbidities (assessed by the clinician at screening only
* BMI>40
* Presence of an acute disease process that might interfere with test performance
* Subjects with PPG SNR <100 indicated by the CardiacSense1 device
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | 24 hours
  Capnograph and Cardiacsense1 sensor Respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Giris Jacob, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD to be shared with other researcher